CLINICAL TRIAL: NCT00522405
Title: Randomized Control Trial (RCT) of Transarterial Chemoembolization (TACE) Versus TACE and Oral Drug Therapy in the Treatment of Unresectable Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-39/29.1.2007; ICMR No-5/8/7/26/99-ECD-I
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2007-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Transarterial chemoembolisation; Thalidomide; Capecitabine; Treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Transarterial Chemoembolisation
  Interventions: Procedure: TACE
- 2 (Active Comparator): TACE Plus oral chemotherapy
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — * Under local anesthesia, the Femoral artery would be punctured
  * A catheter would be introduced and a flush aortogram, superior mesenteric arterioportography and the celiac artery run would be undertaken to define the size and location of the tumors, feeding vessels and to assess the portal vein patency
  * Superselective catheterization of the hepatic artery feeding the tumor would be done
  * By placing the catheter tip beyond the gastroduodenal artery, the chemotherapeutic drugs would be administered.
  * Stable drug mixture would be prepared by using Doxorubicin 50mg, Cisplatin 100mg in combination with 10-15ml of ionic contrast media and 10-20ml of lipiodol by continuously agitating the mixture.
  * The drug mixture would then be injected through the indwelling arterial catheter by continuously flushing alternately, repeatedly and rapidly between two-luer locks syringes connected across a three way.
  * Gelfoam particles would be injected following this for embolization

SUMMARY:
Background Hepatocellular carcinoma, a malignant tumor of liver is one of the most common cancers worldwide. All India Institute Of Medical Sciences (AIIMS) being a tertiary care hospital receives about two to three cases of Hepatocellular carcinoma (HCC) each day in our Gastroenterology out patient department. Most of these patients present late when the disease is already advanced and no curative therapies can be offered. At this stage, palliative therapy forms the mainstay of treatment. This includes TACE or Oral chemotherapy. Whether oral chemotherapy administered along with TACE potentiates the effect and further prolongs survival, needs to be ascertained. No studies of this kind are available.

This prospective study is therefore designed to address this issue.

DETAILED DESCRIPTION:
1. Subjects Consecutive patients of unresectable HCC diagnosed from January 2006 at the liver clinic, AIIMS will be included in the study if they fulfill the following criteria-

   Inclusion criteria · Patients above 12 years of age with performance status (PST)score of 0-2

   · Unresectable HCC with underlying Child's A/B cirrhosis

   · Normal Main portal vein and its branches
   * Normal Inferior vena cava
   * No history of drug allergy
   * Informed written consent of patient.
   * Less than 50% involvement of liver by HCC

   Exclusión criteria

   · Unresectable HCC with underlying Child's C cirrhosis

   · Performance status 3-5

   · Extrahepatic disease

   · Vascular involvement
   * Co-morbid illness like coronary artery disease, congestive heart failure, chronic renal failure etc
   * Previous history of encephalopathy/ upper gastrointestinal bleed in the last six months
   * HCC in a female of child bearing age
2. Diagnostic criteria

   * Cirrhosis of liver- Diagnosis will be founded on the basis of clinical, biochemical and endoscopy findings.
   * Hepatocellular carcinoma- when any one of the following is present

<!-- -->

1. Any two imaging modalities(Ultrasound (US), dual phase CT (DPCT)/ contrast enhanced MRI) showing arterialization of the hepatic mass
2. AFP more than 400ng/ml along with arterialisation on one imaging modality (DPCT/ contrast enhanced MRI)
3. FNAC

3. Randomization

· Patients will be randomized after the confirmation of diagnosis and obtaining written consent

· Sequences will be generated by the Statistician

· Stratified randomization will be done. Two strata of child's A and B will be made

· Randomization will be done by drawing consecutively numbered opaque sealed envelopes

· Randomization into A (TACE) and B (TACE +oral chemotherapy) will be done.

4. Definitions

1. Unresectable HCC-

   · Liver mass larger than 5cm in diameter (single/ multiple), involving less than 50% of the liver.

   · Multiple masses more than three in number and more than 3cm in diameter.
2. Tumor response

   This will be based on Dual phase CT findings

   · Complete response (CR)- Tumor fully covered with lipiodol showing no viable tissue
   * Partial response (PR)- Tumor partially covered (>75%) by lipiodol
   * Mild response (MR)- About 50 to 75% coverage of the tumor by lipiodol
   * No response (NR) - About 25 to 50% coverage of the tumor by lipiodol
   * Fresh lesions (FL)- Appearance of new mass lesions in the liver with or without recurrence at the site of previous mass
3. Patient tolerance- Grade 1: no side effects Grade 2: moderate side effects Grade 3: severe side effects Grade 4: life threatening side effects
4. Performance status (PST score)

   PST score of 0-5 would be assessed on the following basis 0- No cancer related symptoms. Normal life style 1- Minor symptoms related to cancer. Capable of non-strenuous activity. Fully ambulatory 2- Ambulatory and capable of all self care but unable to carry out any work activities Confined to bed less than 50% of waking hours 3- Capable of only limited self care. Confined to bed more than 50% of waking hours.

   4- Completely disabled. Cannot carry on any self care. Totally confined to bed. 5- Death

   5. Sample Size Systematic review of RCTs for TACE show a 2 year survival of 37%. Expecting that addition of oral drugs would increase survival to 37 to 60%, for a power of 80% and error of 5%, a sample size of 73 patients in each arm would be required (Total 146 patients).

   6. Procedure of TACE

   · Patient would be admitted a day prior to the procedure

   · Patient would be made to fast overnight with intravenous fluid infusion started for maintaining hydration

   · Pre-procedure analgesic (3rd generation antibiotic) would be started at a dose of 2gm intravenously, 12 hourly, at least 12 hour before the procedure and continued 5 days post procedure

   · Under local anesthesia, the Femoral artery would be punctured at the upper thigh with a Medicut 18 gauge

   · A catheter would be introduced through this route with the help of a guide wire and a flush aortogram, superior mesenteric arterioportography and the celiac artery run would be undertaken to define the size and location of the tumors, feeding vessels and to assess the portal vein patency

   · Superselective catheterization of the hepatic artery feeding the tumor would be done

   · By placing the catheter tip beyond the gastroduodenal artery, the chemotherapeutic drugs would be administered.

   · Stable drug mixture would be prepared by using Doxorubicin 50mg, Cisplatin 100mg in combination with 10-15ml of ionic contrast media and 10-20ml of lipiodol by continuously agitating the mixture.

   · Hydrocortisone 100mg and augmenting dose of analgesic and sedative would be injected prior to the administration of the drug.

   · The drug mixture would then be injected through the indwelling arterial catheter by continuously flushing alternately, repeatedly and rapidly between two lever lock syringes connected across a three way.

   · Gelfoam particles would be injected following this for embolization

   · Post procedure, devascularization would be confirmed by additional angiography of the hepatic artery.

   · Procedure would last approx 45mts-1 hour.

   · Tight compression would be given at the punctured site and patient would be shifted to the ward once complete hemostasis is achieved.

   7. Follow up post TACE Clinical follow up
   * All patients would be followed up in the Liver clinic monthly unless their clinical condition warrants earlier follow up
   * Liver function tests/ complete blood count would also be done at each visit and AFP (if elevated earlier) every six months
   * Patient tolerance, child's status would be estimated. Imaging follow up
   * At one month, a dual phase CT would be done to ascertain the response to therapy and the need to repeat the procedure. Subsequently, the DPCT would be done at 3 and 6 monthly intervals.
   * Once the tumor shows complete coverage, randomization into the two treatment groups would be done

     9. Repeat TACE on follow up This would be done if any of the following is noted
   * DPCT shows viable tumor
   * Fresh lesions appear
   * Elevated serum AFP occurs with or without appearance of viable mass on DPCT

     10. Oral chemotherapy Drugs used would be Thalidomide and Capecitabine in the following dosage schedule-

   Thalidomide---100mg once a day (OD) for 7 days, Increased to 200mg OD for 7 days, further increased to 300mgOD for 7 days till a maximum of 600mg once a day is reached

   Capecitabine---- 500mg OD for 7 days, then 1000mg OD for next 7 days, increased to a maximum dose of 1500mg OD.

   Total leucocyte count & Platelet count would be monitored every 15 days

   11. Duration of follow up- Two years after achieving total coverage of the mass lesion on DPCT

   12. Outcome measures Following parameters will be used to ascertain the outcome of treatment
   1. Primary Outcome

      1. Survival rate- calculated from the start of TACE
      2. End point Group 1 - Progression of disease and repeat TACE is not possible Group 2 - Death
   2. Secondary Outcome

      1. Tumor response on dual phase CECT
      2. Patient tolerance
      3. Childs' status of cirrhosis- will be ascertained at one and two years of follow up depending upon the Childs' scoreScore <6- Childs'A, 7-9 Childs'B and >10 Childs'C

ELIGIBILITY:
Inclusion Criteria:

* Patients above 12 years of age with performance status (PST)score of 0-2
* Unresectable HCC with underlying Child's A/B cirrhosis
* Normal Main portal vein and its branches
* Normal Inferior vena cava
* No history of drug allergy
* Informed written consent of patient.
* Less than 50% involvement of liver by HCC

Exclusion Criteria:

* Unresectable HCC with underlying Child's C cirrhosis
* Performance status 3-5
* Extrahepatic disease
* Vascular involvement
* Co-morbid illness like coronary artery disease, congestive heart failure, chronic renal failure etc
* Previous history of encephalopathy/ upper gastrointestinal bleed in the last six months
* HCC in a female of child bearing age

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Survival rate- calculated from the start of TACE

SECONDARY OUTCOMES:
a) Tumor response on dual phase CECT b) Patient tolerance c) Childs' status of cirrhosis- will be ascertained at one and two years of follow up depending upon the Childs' scoreScore <6- Childs'A, 7-9 Childs'B and >10 Childs'C

CONTACTS AND LOCATIONS:
Overall Officials: Subrat K Acharya, DM, Principal Investigator — All India Institute of Medical Sciences, New Delhi, India
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- See also: All India Institute of Medical Sciences, New Delhi, India — http://www.aiims.edu